CLINICAL TRIAL: NCT03358485
Title: A Single-center, Randomized, Doule Blind, Placebo-controlled, Multiple Dose Escalation Phase 1b Study to Evaluate the Safety and Tolerability of Aolanti Weikang Tablets in Healthy Volunteers
Brief Title: Study of Aolanti Weikang Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QF-WKP-101
Record Dates: First submitted 2017-11-27; First posted 2017-11-30 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2017-12

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aolanti Weikang tablets (Experimental): 3，6 or 8 Aolanti Weikang tablets each time,tid
  Interventions: Drug: Aolanti Weikang tablets
- Placebo (Placebo Comparator): 3,6 or 8 tablets each time,tid
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aolanti Weikang tablets — Aolanti Weikang tablets is a Chinese patent drug designed to treat Functional dyspepsia (FD).
  Arms: Aolanti Weikang tablets
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple doses escalation of Aolanti Weikang tablets to determine the MTD in healthy volunteers

DETAILED DESCRIPTION:
This is a single-center, randomized, doule blind, placebo-controlled, multiple dose escalaction phase 1b study to evaluate the safety and tolerability of Aolanti Weikang tablets in healthy volunteers. Aolanti Weikang tablets is a Chinese patent drug designed to treat Functional dyspepsia (FD). The proposed dose escalaction levels is 3,6 and 8 tablets. If MTD is not established up to 8 tablets, the dose escalaction will be stopped. In each dose level, subjects will be randomly given orally Aolanti Weikang tablets or placebo tablets at a 3:1 ratio three times a day (tid) for 7 consecutive days, then will receive the Safety follow up for 14 days. No intrapatient dose-escalation is permitted.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) :≥19 and ≤26 kg/m2
* Signed written informed consent

Exclusion Criteria:

* With in 7 days of Screening, the average number of stool > 2 times/day
* With in 7 days of Screening, with the presence of ≥ type 5 stool form per the Bristol Stool Form Scale
* At least one clinically significant abnormality based the comprehensive examination (including vital signs, physical examination, laboratory examination and others)
* Digestive diseases, or other diseases within 3 months that may affect the swallow, absorption, or metabolism of study drugs, and not yet fully recovered judged by the Investigator
* Smoking, alcohol abuse or drug abuse with in 3 months or drinking within 48 hours before the first administration
* History of drug or aurantium allergy
* Concomitant medication within 2 weeks prior to drug administration or any drug being used
* Participated in other clinical trials within 3 months before Screening
* Major surgery/surgical therapy for any cause within 4 weeks of Screening, or scheduled surgeries within 2 weeks after the last dose of study drug
* Subjects not agree to use adequate contraception from study entry through at least 28 days after the last dose of study drug
* Pregnancy or nursing
* Other conditions that unsuitable for enrollment considered by Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated Dose (MTD) of Aolanti Weikang tablets | 3 weeks
  Definition of MTD: the dose level at which 3 or more subjects experienced one or more dose limited toxicities

SECONDARY OUTCOMES:
Number and grade of treatment-related adverse events (AEs) | 3 weeks
  All of the AE are assessed by NCI-CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Tang, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No